CLINICAL TRIAL: NCT03690349
Title: Is Mold Sensitization Associated With Severe Asthma Exacerbation in Children?
Brief Title: Mold Sensitization Associated Severe Asthma Exacerbation
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: 271/2560(EC4)
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: severe asthma exacerbation; Mold sensitization
MeSH Terms: conditions — Asthma | interventions — Skin Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skin test in severe asthma exacerbation: Skin test in asthmatic children hospitalized due to severe asthma exacerbation in a preceding year
  Interventions: Other: Skin test
- skin test in outpatient: Skin test in asthmatic children without severe asthma exacerbation in a preceding year
  Interventions: Other: Skin test

INTERVENTIONS:
Other: Skin test — Demographic data review, Disease severity evaluation, Treatment evaluation and Skin prick test for 16 common aeroallergens

SUMMARY:
Mold sensitization is associated with severe asthma exacerbation.

DETAILED DESCRIPTION:
Mold sensitization has been reported to be one of the factors that is associated with severe asthma exacerbation (SAE). The objective is to identify the factors that are associated with SAE in asthmatic children particularly mold sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic children aged 1-15 years old from Pediatric Allergy and Immunology division with hospitalized due to severe asthma exacerbation in a preceding year and without severe asthma exacerbation in a preceding year

Exclusion Criteria:

* Other serious systemic diseases, pregnant, lactation

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthmatic children aged 1-15 years old from Pediatric Allergy and Immunology division devided in to 2 groups: 1. hospitalized due to severe asthma exacerbation in a preceding year and 2. without severe asthma exacerbation in a preceding year
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Association between mold sensitization and severe asthma exacerbation | 1 year
  Compare mean wheal diameter (mm.) of skin prick test of mold allergen extracts between the group with severe asthma exacerbation and the group without severe asthma exacerbation

IPD SHARING:
Plan to Share IPD: Undecided